CLINICAL TRIAL: NCT01654107
Title: Persistence-Targeted Smoking Cessation
Acronym: PTSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220110199; R34DA030652 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco; smoking cessation; nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Persistence Targeted Smoking Cessation (Experimental): Persistence Targeted Smoking Cessation - 8 weeks counseling + 12 weeks nicotine lozenge
  Interventions: Behavioral: Persistence Targeted Smoking Cessation; Drug: Nicotine lozenge
- Clearing The Air (Active Comparator): Clearing the Air Smoking Cessation intervention - 8 weeks counseling + 12 weeks nicotine lozenge
  Interventions: Behavioral: Clearing The Air; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Persistence Targeted Smoking Cessation — 8-weeks of smoking cessation counseling ("Persistence Targeted Smoking Cessation")
  Other Names: PTSC
  Arms: Persistence Targeted Smoking Cessation
Behavioral: Clearing The Air — 8-weeks counseling + 12-weeks nicotine lozenge based on NCI protocol, Clearing The Air
  Other Names: CTA
  Arms: Clearing The Air
Drug: Nicotine lozenge — 12-weeks 4mg nicotine lozenge

SUMMARY:
The investigators propose to develop a theory-based smoking cessation intervention (called Persistence-targeted smoking cessation; PTSC). PTSC includes 8 weekly individual counseling sessions and use of nicotine lozenge for 12 weeks. The investigators will test the feasibility and preliminary efficacy of the intervention (i.e., cigarettes per day and prolonged abstinence).

DETAILED DESCRIPTION:
In this Stage I Behavioral & Integrative Treatment Development (R34) project, we propose to develop a theory-based smoking cessation intervention (called Persistence-targeted smoking cessation; PTSC). PTSC includes 8 weekly individual counseling sessions and use of nicotine lozenge for 12 weeks. We will test the feasibility and preliminary efficacy of the intervention (i.e., cigarettes per day and prolonged abstinence). We hope to develop a feasible psychosocial treatment for use in a later randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 - 64 years old
* Must smoke at least 10 cigarettes per day for past 6-months
* Expired breath carbon monoxide (CO) > 7
* Must have a working cellular phone

Exclusion Criteria:

* Must not be currently receiving tobacco dependence treatment counseling
* Must not currently be taking varenicline, bupropion, or any nicotine preparations (gum, lozenge, patch, spray, inhaler)
* Must have no contraindications to using nicotine lozenge

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Steinberg, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Persistence Targeted Smoking Cessation | Clearing The Air
Started | 28 | 30
Completed | 25 | 22
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Persistence Targeted Smoking Cessation | Clearing The Air | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.82 (10.205) | 48.93 (8.574) | 48.40 (9.330)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Abstinence
Description: 3-months after the Quit Date
Time Frame: 3-months
Measure: Number; unit: participants
Arm/Group | Persistence Targeted Smoking Cessation | Clearing The Air
Number analyzed (Participants) | 25 | 28
participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Persistence Targeted Smoking Cessation | Clearing The Air
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 19/28 | 13/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Persistence Targeted Smoking Cessation (N=28) | Clearing The Air (N=30)
Dry Mouth (General disorders) | 1 | 2
Throat irritation (General disorders) | 8 | 4
Upset stomach (Gastrointestinal disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Heartburn (Gastrointestinal disorders) | 2 | 0
Hiccups (General disorders) | 4 | 0
Coughing (General disorders) | 2 | 1
Sore throat (General disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Cold symptoms (Immune system disorders) | 1 | 2
Decreased appetite (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Nasal congestion (Immune system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Tooth ache (General disorders) | 1 | 0
Irregular Bowel Movement (Gastrointestinal disorders) | 1 | 0
Heart flutter (Cardiac disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Sweating (General disorders) | 0 | 1
Nose flaring (General disorders) | 0 | 1
Burning sensation in cheek area (General disorders) | 0 | 1
Sore gums (General disorders) | 0 | 1
Canker sore (General disorders) | 0 | 1
Gas (Gastrointestinal disorders) | 0 | 1
Fibromyalgia pain worsening (Nervous system disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 2
Poor concentration/forgetfulness (Psychiatric disorders) | 0 | 1
Increased appetite (Gastrointestinal disorders) | 0 | 1
Burning pepper taste (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No